CLINICAL TRIAL: NCT00125073
Title: Postoperative Dietary Counseling After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK67885; R03DK067885 (NIH)
Record Dates: First submitted 2005-07-28; First posted 2005-07-29 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Obesity
Keywords: Standard Care; Nutritional Counseling
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: Postoperative nutritional counseling

SUMMARY:
This study aims to assess the changes in physical characteristics, food intake, eating behavior, vomiting, and dumping in 100 patients who undergo bariatric surgery. Patients are put into one of two conditions; they will either receive standard postoperative care or biweekly counseling sessions with a dietician that will help them with the postoperative diet. Patients who receive dietary counseling are anticipated to experience greater weight loss and report less consumption of sugar and fat as compared to patients who do not receive dietary counseling. Moreover, patients who receive dietary counseling are predicted to report less frequent nausea, vomiting, and gastric dumping, as compared to patients who do not receive postoperative dietary counseling. This is predicted to result as a consequence of increased dietary adherence evidenced by the former group.

DETAILED DESCRIPTION:
This study aims to assess the changes in physical characteristics, food intake, eating behavior, vomiting, and dumping in 100 patients who undergo bariatric surgery. Patients are put into one of two conditions; they will either receive standard postoperative care or biweekly counseling sessions with a dietician that will help them with the postoperative diet. Patients who receive dietary counseling are anticipated to experience greater weight loss and report less consumption of sugar and fat as compared to patients who do not receive dietary counseling. Moreover, patients who receive dietary counseling are predicted to report less frequent nausea, vomiting, and gastric dumping, as compared to patients who do not receive postoperative dietary counseling. This is predicted to result as a consequence of increased dietary adherence evidenced by the former group.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): 40 to 60 kg(squared) or greater than or equal to 35kg(squared) in the presence of co-morbid medical condition.
* Subjects must live within 30 minutes of the University of Pennsylvania and drive or have ready access to public transportation.
* Subjects must be able to ambulate without assistance.
* Subjects will be free of contraindications to bariatric surgery and will have been approved for surgery by both the medical staff and their insurance carrier.
* Subjects must be able to communicate with the investigator, be legally competent, and provide written informed consent.

Exclusion Criteria:

* Evidence of significant psychiatric distress that impairs daily functioning, as suggested by a Beck Depression Inventory-II (BDI-II) greater than or equal to 25. (Individuals with BDI-II scores greater than or equal to 25 will be referred for appropriate help, as per the requirements of the law in the state of Pennsylvania.)
* Any current substance abuse or dependence disorder.
* Concurrent psychiatric treatment for any DSM-IV condition
* Persons who binge eat and report purging behavior (i.e., vomiting, laxative or diuretic abuse, etc.) will be excluded from the study and referred to an eating disorders specialist.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-07; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Sarwer, Ph.D., Principal Investigator — The University of Pennsylvania
Locations (1):
- The University of Pennsylvania Weight and Eating Disorder Program, Philadelphia, Pennsylvania, United States